CLINICAL TRIAL: NCT05240690
Title: Clinical Study on the Safety and Efficacy of Umbilical Cord Blood Derived MAK Immune Cells Combined With Standard Second-Line Treatments for Hepatobiliary and Pancreatic Malignancies：HCCSC AB04 Trial
Brief Title: Umbilical Cord Blood Derived MAK Immune Cells Combined With Standard Second-Line Treatments for Hepatobiliary and Pancreatic Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhou Fuxiang (Other)
Responsible Party: Sponsor-Investigator, Zhou Fuxiang, Professor, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC AB04
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Stage IV Pancreatic Cancer; Hepatocellular Carcinoma , Cholangiocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Umbilical Cord Blood Derived MAK Immune Cells (Experimental)
  Interventions: Biological: Umbilical Cord Blood Derived MAK Immune Cells

INTERVENTIONS:
Biological: Umbilical Cord Blood Derived MAK Immune Cells — Intravenous drip
  Other Names: Second-line standard treatment

SUMMARY:
To evaluate the safety of MAK immune cells derived from umbilical cord blood combined with second-line treatments for hepatobiliary and pancreatic malignancies.And to investigate the initial efficacy of MAK immune cells derived from umbilical cord blood combined with second-line treatments for hepatobiliary and pancreatic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old, under 75 years old, men and women;
2. Subjects participated voluntarily, gave full informed consent, signed a written informed consent, with good compliance;
3. Hepatocytic carcinoma or biliary or pancreatic-derived adenocarcinoma was clearly diagnosed by histological or cytology pathology;
4. Recurrent hepatobiliary or pancreatic malignancies with unresectable advanced or metastatic, or postoperative adjuvant therapy (chemotherapy and / or radiation therapy) for 12 months, with a Child-Pugh score of 7;
5. With 1 measurable lesion, according to the RECIST v 1.1 criteria.Requirements: The selected target lesion has not previously received local treatment, or the selected target lesion was located in the previous local treatment area after passing the imaging examination and was determined as PD according to the RECIST v 1.1 criteria;
6. ECOG score of 0-1;
7. Expected survival is greater than 3 months;
8. Main organ function composite with the following requirements:

   * Absolute neutrophil count was 1.5*10^9 / L;
   * Platelet count was 75*10^9 / L;
   * Hemoglobin was at 90g / L;
   * Serum albumin at 30g / L;
   * Serum bilirubin 1.5 upper Range normal limit (ULN);
   * Altraverine aminotransferase (ALT), aspartate aminotransferase (AST) 2.5 upper normal range limit (ULN);
   * Serum creatinine (Cr) 1.5 Upper Limit of normal range (ULN) or Cr clearance of 40 mL/min;
   * The International standardized ratio (INR) 2 or Prothrombin Time (PT) exceeds the upper limit of the normal range for 6 seconds;
   * Urinary protein <2 + (if urine protein 2 +, 24 h (h), and 24h <1.0g can be enrolled).

     9.If HBsAg (+) and / or HBcAb (+), HBV DNA must be <500IU / mL and during the study period, the original anti-HBV treatment continues throughout the study, or start entecavir or teenofavir.

     10.There is no previous history of abdominal radiotherapy. If radiation has been performed, the complete target area scope and treatment plan are more than 2 weeks apart from the study immune cell transfusion of this project; 11.No history of organ transplantation; 12.Women of childbearing age performed a serum pregnancy test within 7 days before the initiation of treatment, and agreed to adopt a reliable and effective contraceptive method during the trial and within 60 days after the final administration of the test drug.For male subjects with a partner of women of childbearing age, consent was given to a reliable and effective approach to contraception during the trial and within 60 days after the final administration of the test medication.

Exclusion Criteria:

1. At the same time, there are serious medical diseases, including serious heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled infection, active digestive tract ulcer;
2. Patients with brain metastasis with clinical symptoms;
3. Suffering from other primary malignancies in the past 5 years (except skin BCC or squamous cell carcinoma, cervical carcinoma in situ that have been effectively controlled);
4. Patients with immunodeficiency or autoimmune diseases (e. g., rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, insulin-dependent diabetes, etc.).
5. Patients who participated in other clinical trials or clinical study treatment within the 3 months prior to this clinical study.
6. Patients treated with other cells within the last 6 months.
7. Patients with infection and fever who were not effectively controlled.
8. Patients with high allergies or a history of severe allergies.
9. Patients with an albumin allergy.
10. Patients after organ transplantation; patients with long-term use or who are using immunosuppressants.
11. Patients with severe other organ dysfunction.
12. Patients with organ bleeding, severe hypertension, and patients with a cardiac pacemaker.
13. Women during pregnancy or lactation; or women of childbearing age have positive blood pregnancy, women of childbearing age and their spouses are unwilling to take effective contraception during the clinical study and within 6 months of the end.
14. Patients who are not considered appropriate to participate in this clinical study (e. g., poor compliance, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-02-07 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival(PFS) | 24 months
  PFS is defined as the time from enrollment to the first documented disea

SECONDARY OUTCOMES:
overall survival (OS) | 24 months
  OS is the time from enrollment to death due to any cause.
objective response rate (ORR) | 24 months
  and partial response (PR) by the investigator according to the RECIST 1.1.
disease control rate (DCR) | 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No